CLINICAL TRIAL: NCT05083520
Title: Incidence of Cereblon in Intensive Care Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Buca Seyfi Demirsoy State Hospital (Other)
Responsible Party: Principal Investigator, Pınar Ayvat, Head of Anesthesia and Reanimation Department, Buca Seyfi Demirsoy State Hospital
Other Study IDs: Cereblon
Record Dates: First submitted 2021-09-24; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Critical Illness; Sepsis
Keywords: Critical care; Cereblon
MeSH Terms: conditions — Critical Illness; Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critical care patients

SUMMARY:
Classical immunomodulatory drugs (IMiDs) like thalidomide and its second- and third-generation analogues lenalidomide, pomalidomide, avadomide (CC-122), and iberdomide (CC-220) have constantly emerged to new therapeutic areas. Originally developed as a sedative and banned in 1961 for its teratogenic effects when used during pregnancy, thalidomide and a number of newly developed analogues are approved for the treatment of multiple myeloma (MM),4 erythema nodosum5 and myelodysplastic syndrome (MDS) Thalidomide was used as a treatment for morning sickness from 1957 until 1961 but was withdrawn from the market after it was discovered that it caused birth defects. Because of their pleiotropic and especially anti-angiogenic properties, IMiDs have further been reported effective in many off-label indications as for Hodgkin's lymphoma, light chain-associated (AL) amyloidosis, and acute myeloid leukemia (AML).

The drug thalidomide binds to cereblon and changes which substrates can be degraded by it, which leads to an antiproliferative effect on myeloma cells and possibly the teratogenic effect on fetal development. The idea that cereblon modulation is responsible for the teratogenic activity of thalidomide in the chick and zebrafish was cast into doubt due to a 2013 report that pomalidomide (a more potent thalidomide analog) does not cause teratogenic effects in these same model systems even though it binds with cereblon more strongly than thalidomide.

Cereblon (CRBN) is a substrate receptor of the E3 ubiquitin ligase complex. Several key findings suggest diverse roles of CRBN, including its regulation of the large-conductance calcium- and voltage-activated potassium (BKCa) channels, regulation of thalidomide-binding proteins, and mediation of lenalidomide treatment in multiple myeloma. Recent studies also indicate that CRBN is involved in energy metabolism and negatively regulates AMP-activated protein kinase signaling. Recent studies also indicate that CRBN is involved in energy metabolism and negatively regulates AMP-activated protein kinase signaling. Mice with genetic depletion of CRBN are resistant to various stress conditions including a high-fat diet, endoplasmic reticulum stress, ischemia/reperfusion injury, and alcohol-related liver damage.

There are different drugs that have an immunomodulating effect, such as thalidomide analogs, and are used in various situations. Some of the diseases in which the immune system plays a role in its etiology are Acute Respiratory Distress Syndrome (ARDS), Acute Lung Injury (ALI), septic shock, and sepsis. In cases of lung injury such as sepsis, septic shock, ARDS, ALI, the immune system is over-activated and as a result, the immune system cells damage the own tissue of the lung. To break this mechanism, immunomodulatory drugs are used in intensive care in the treatment of these diseases.

There is no publication regarding the role of Cereblon in the mechanism of action of these immunomodulatory drugs used in intensive care. In these intensive care diagnoses (sepsis, ARDS, ALI), there is no publication showing the correlation between the severity of the disease and Cereblon protein. Other laboratory parameters are used to estimate the effects (mortality and morbidity) of these diseases on the patient. At the end of the investigators study, the investigators think that the Cereblon gene can be used in this estimation of mortality or morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Having (-) Covid PCR test,
* Being intubated,
* Getting permission from the patient's relatives to be included in the study

Exclusion Criteria:

* Being under the age of 18,
* Having (+) Covid PCR test,
* Not be able to get consent from the relatives of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critical care patient
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
The presence of Cereblon protein | until 31 December 2021
  To demonstrate the presence of Cereblon protein in tracheal aspiration fluid from intensive care patients.

SECONDARY OUTCOMES:
The relationship between Cereblon and intensive care length of stay | until 31 December 2021
  To determine whether there is a relationship between the presence of Cereblon protein and the length of stay in the intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Ayvat, ass. prof., Study Chair — Izmir Democracy University

REFERENCES:
- [Background] Yang H, Song Z, Hong D. CRBN knockdown mitigates lipopolysaccharide-induced acute lung injury by suppression of oxidative stress and endoplasmic reticulum (ER) stress associated NF-kappaB signaling. Biomed Pharmacother. 2020 Mar;123:109761. doi: 10.1016/j.biopha.2019.109761. Epub 2019 Dec 19. PMID 31865141
- [Background] Gil M, Kim YK, Kim HY, Pak HK, Park CS, Lee KJ. Cereblon deficiency confers resistance against polymicrobial sepsis by the activation of AMP activated protein kinase and heme-oxygenase-1. Biochem Biophys Res Commun. 2018 Jan 1;495(1):976-981. doi: 10.1016/j.bbrc.2017.11.098. Epub 2017 Nov 21. PMID 29170136